CLINICAL TRIAL: NCT01386970
Title: Sex and Disease Dependent Nucleoside Analog Toxicity
Brief Title: Effect of Gender and HIV Infection on Zidovudine and Lamivudine Pharmacokinetics
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); University of Hawaii (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 04-1101; R01AI064029 (NIH)
Record Dates: First submitted 2011-06-28; First posted 2011-07-01 (Estimated); Results first posted 2020-03-16 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: HIV
Keywords: Pharmacokinetics; antiretroviral therapy; nucleoside analogs; mitochondrial toxicity; clinical pharmacology; cellular pharmacology; pharmacogenetics
MeSH Terms: interventions — Zidovudine; Lamivudine; lamivudine, zidovudine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HIV-negative (Active Comparator): This group was used to compare intracellular ZDV- and 3TC-triphosphate concentrations to the HIV-infected group and in men versus women.
  Interventions: Drug: zidovudine 300mg and lamivudine 150mg as Combivir
- HIV-infected (Active Comparator): This group was started on ZDV-3TC based therapy. Intracellular ZDV- and 3TC-triphosphate concentrations were compared in men versus women and the HIV-negative group.
  Interventions: Drug: zidovudine 300mg and lamivudine 150mg as Combivir

INTERVENTIONS:
Drug: zidovudine 300mg and lamivudine 150mg as Combivir — twice daily for 12 days in the HIV-negative group and indefinitely for their care in the HIV-positive group

SUMMARY:
This study evaluated the blood and blood cell concentrations of zidovudine and lamivudine in men versus women and in those with versus without HIV infection. Additionally, markers of side effects were correlated with blood levels of the drugs. The hypothesis was that women and those with HIV would have higher drug levels, as well as markers of side effects.

ELIGIBILITY:
Inclusion Criteria:

* Documented physician-diagnosed HIV-infection (HIV+ antibody or plasma HIV-RNA+); HIV-negative volunteers must have a negative HIV-ELISA.
* Age 18 to 55 years;
* Either antiretroviral naïve, or no HIV-therapy in the preceding 6 months;
* Planned antiretroviral regimen includes standard doses of ZDV plus 3TC as part of the antiretroviral regimen. Once- or twice-daily 3TC will be allowed.

Exclusion Criteria:

* Any medical condition that in the opinion of the investigators would jeopardize the intent of the study.
* In the opinion of the investigator, any concomitant immunomodulatory medications, chemotherapeutic agents, investigational drugs, and alternative therapies, including, glucocorticoids, recombinant growth factors or cytokines (e.g. Granulocyte-macrophage colony-stimulating factor, Granulocyte colony-stimulating factor, interferon-alpha or gamma, human growth hormone, etc), ribavirin, birth-control pills, and sex hormones that could interfere with the cellular pharmacology of the study medications;
* Concomitant medications that interfere with renal drug clearances including, tenofovir, adefovir, cidofovir, ganciclovir, probenecid, or any similarly problematic medication in the opinion of the investigators;
* Concomitant warfarin or daily aspirin (to prevent excess bleeding from biopsy).
* Pregnancy or a plan to become pregnant, or menopause;
* Any > or = grade II abnormality in hemoglobin, absolute neutrophil count, routine liver function tests, serum creatinine, or other organ function abnormalities.
* Any medical or personal condition that, in the judgment of the investigators, may influence the subject's ability to comply with study conditions, such as active mental illnesses, or plans to leave the geographical area.
* Inability to give informed consent.
* Triple nucleoside analog reverse transcriptase regimens.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2005-05; Primary Completion 2008-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter L. Anderson, PharmD, Principal Investigator — University of Colorado Denver and Health Sciences Center
Locations (1):
- University of Colorado Denver and Health Sciences Center, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share.

REFERENCES:
- [Background] Anderson PL. Recent developments in the clinical pharmacology of anti-HIV nucleoside analogs. Curr Opin HIV AIDS. 2008 May;3(3):258-65. doi: 10.1097/COH.0b013e3282f85dc1. PMID 19372976
- [Background] Anderson PL, Rower JE. Zidovudine and Lamivudine for HIV Infection. Clin Med Rev Ther. 2010;2:a2004. PMID 20953318
- [Background] Ghodke Y, Anderson PL, Sangkuhl K, Lamba J, Altman RB, Klein TE. PharmGKB summary: zidovudine pathway. Pharmacogenet Genomics. 2012 Dec;22(12):891-4. doi: 10.1097/FPC.0b013e32835879a8. No abstract available. PMID 22960662
- [Result] Rower JE, Klein B, Bushman LR, Anderson PL. Validation of a sensitive LC/MS/MS method for the determination of zidovudine and lamivudine in human plasma. Biomed Chromatogr. 2012 Jan;26(1):12-20. doi: 10.1002/bmc.1617. Epub 2011 Apr 4. PMID 21465499
- [Result] Anderson PL, Zheng JH, King T, Bushman LR, Predhomme J, Meditz A, Gerber J, Fletcher CV. Concentrations of zidovudine- and lamivudine-triphosphate according to cell type in HIV-seronegative adults. AIDS. 2007 Sep 12;21(14):1849-54. doi: 10.1097/QAD.0b013e3282741feb. PMID 17721092
- [Result] Rower JE, Meditz A, Gardner EM, Lichtenstein K, Predhomme J, Bushman LR, Klein B, Zheng JH, Mawhinney S, Anderson PL. Effect of HIV-1 infection and sex on the cellular pharmacology of the antiretroviral drugs zidovudine and lamivudine. Antimicrob Agents Chemother. 2012 Jun;56(6):3011-9. doi: 10.1128/AAC.06337-11. Epub 2012 Mar 5. PMID 22391541

RESULTS

PARTICIPANT FLOW:
Groups:
- HIV-negative: This group was used to compare intracellular ZDV- and 3TC-triphosphate concentrations to the HIV-infected group and in men versus women.
  zidovudine 300mg and lamivudine 150mg as Combivir: twice daily for 12 days in the HIV-negative group
- HIV-infected: This group was started on ZDV-3TC based therapy. Intracellular ZDV- and 3TC-triphosphate concentrations were compared in men versus women and the HIV-negative group.
  zidovudine 300mg and lamivudine 150mg as Combivir: indefinitely for their care in the HIV-positive group
Period: Overall Study
Arm/Group | HIV-negative | HIV-infected
Started | 20 | 23
Completed | 16 | 21
Not Completed | 4 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Adverse Event | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HIV-negative | HIV-infected | Total
Number analyzed (Participants) | 20 | 23 | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 23 | 43
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 12 | 17 | 29
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 4 | 7 | 11
  Non- African-American | 16 | 16 | 32

OUTCOME MEASURES:

1. Primary Outcome: ZDV-TP Drug Levels Compared Between HIV Negative and HIV Infected Subject
Description: To compare ZDV- triphosphate concentrations in HIV-negative versus HIV-infected subjects.
Time Frame: Day 12 of dosing
Measure: Median (Inter-Quartile Range); unit: pmol/10^6 cells
Groups:
- HIV-negative; HIV-infected: This group was used to compare intracellular ZDV-triphosphate concentrations to the HIV-infected group
  zidovudine 300mg twice daily for 12 days in the HIV-negative group
Arm/Group | HIV-negative | HIV-infected
Number analyzed (Participants) | 20 | 23
pmol/10^6 cells | 33.89 [28.82 to 42.96] | 29.7 [22.09 to 45.77]

2. Primary Outcome: 3TC-TP Drug Levels Compared Between HIV Negative and HIV Infected Subject
Description: To compare 3TC- triphosphate concentrations in HIV-negative versus HIV-infected subjects.
Time Frame: Day 12 of dosing
Measure: Median (Inter-Quartile Range); unit: pmol/10^6 cells
Groups:
- HIV-negative: This group was used to measure intracellular 3TC-triphosphate concentrations in those who are HIV-negative
  lamivudine 150mg twice daily for 12 days in the HIV-negative group
- HIV-infected: This group was used to measure intracellular 3TC-triphosphate concentrations in those who are HIV-positive
  lamivudine 150mg twice daily indefinitely for their care in the HIV-positive group
Arm/Group | HIV-negative | HIV-infected
Number analyzed (Participants) | 20 | 23
pmol/10^6 cells | 7.25 [6.02 to 8.05] | 5.3 [4.37 to 6.15]

ADVERSE EVENTS:
Time Frame: Time of consenting to study exit (Day 12 or earlier).
Description: AEs were graded per the DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 1.0 - December 2004 (Clarification dated August 2009) (US Dept HHS, NIH, NIAID) Available from: https://rsc.niaid.nih.gov/sites/default/files/table-for-grading-severity-of-adult-pediatric-adverse-events.pdf
Arm/Group | HIV-negative | HIV-infected
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/23
Other Adverse Events (participants affected / at risk) | 7/20 | 8/23
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HIV-negative (N=20) | HIV-infected (N=23)
Abnormal lab- Bilirubin (Hepatobiliary disorders) | 7 | 8 — bilirubin increase
Abnormal Lab- albumin (Hepatobiliary disorders) | 0 | 6 — Decrease in albumin
Abnormal Lab- Alanine Aminotransferase (ALT) (Hepatobiliary disorders) | 0 | 7 — increase in Alanine Aminotransferase (ALT)
Abnormal Lab- Aspartate transaminase (AST) (Hepatobiliary disorders) | 0 | 7 — increase in Aspartate transaminase (AST)
Abnormal Lab- Amylase (Endocrine disorders) | 0 | 7 — Increase in amylase
Nausea, Vomiting, and/or Diarrhea (Gastrointestinal disorders) | 4 | 1 — GI distress leading to subject withdrawal

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No